CLINICAL TRIAL: NCT03382847
Title: A Single-center Pilot Study of the Use of Hepatitis C Positive Donors for Hepatitis C Negative Heart Transplant Recipients With Post-transplant Treatment of Hepatitis C Viremia With Mavyret
Brief Title: HCV Positive Heart Donors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-01775
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): HCV negative patients will receive a heart transplant from a HCV positive donor. Post-transplant, there will be surveillance for the development of viremia, and treatment of viremia. Following treatment, there will be surveillance for a sustained virologic response to HCV treatment.
  Interventions: Combination Product: Transplant with HCV positive donor, followed by surveillance and treatment of viremia

INTERVENTIONS:
Combination Product: Transplant with HCV positive donor, followed by surveillance and treatment of viremia — Heart transplant with HCV positive donor, followed by treatment for viremia if viremia occurs

SUMMARY:
Study subjects active on the waiting list for a heart transplant at the NYU Langone Transplant Institute who are hepatitis C (HCV) negative will receive a heart transplant from a donor who tests positive for HCV. The study will entail surveillance for the development of HCV viremia post-transplant. Patients who develop HCV viremia post-transplant will be treated with an FDA-approved, pan-genotypic direct acting antiviral drug, Mavyret. Patients who are treated with Mavyret will be monitored for clearance of viremia and for sustained virologic response.

ELIGIBILITY:
Inclusion Criteria:

* Listed for an isolated heart transplant at NYU Langone Health
* Able to travel to the NYU Langone Health for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
* No active illicit substance abuse
* Weight at least 50kg
* Women of childbearing potential must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) after transplant due to the increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method after transplant to prevent any secretion exchange
* Able and willing to provide informed consent

Exclusion Criteria:

* HIV positive
* HCV RNA positive or history of previously treated HCV
* Hepatitis B surface antigen positive or on active antiviral treatment for HBV
* Pregnant or nursing (lactating) women
* Use of strong CYP3A inducers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Reyentovich, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Transplant Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 13
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response After Treatment
Description: Percentage of patients with sustained virologic response after treatment for HCV after heart transplant.
Time Frame: 1 year
Population: 100% of surviving patients met this endpoint. One patient expired in the early post-operative period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=25)
pancreatitis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03382847/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03382847/SAP_001.pdf